CLINICAL TRIAL: NCT04572438
Title: COVIDTrach; a UK National Cohort Study of Mechanically Ventilated COVID-19 Patients Undergoing Tracheostomy
Brief Title: A Cohort Study of Mechanically Ventilated COVID-19 Patients Undergoing Tracheostomy
Acronym: COVIDTrach
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: Z6364106/0000/00/00
Record Dates: First submitted 2020-09-29; First posted 2020-10-01 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Tracheostomy Complication; Covid19; Ventilator Lung
MeSH Terms: conditions — COVID-19 | interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tracheostomy — Tracheostomy is a procedure that creates a surgical airway in the windpipe to improve oxygenation of the lungs.

SUMMARY:
COVIDTrach aims to assess the outcomes of tracheostomy in mechanically ventilated patients with COVID-19. The use of personal protective equipment and incidence of COVID-19 amongst operators is also recorded.

DETAILED DESCRIPTION:
COVID-19 can lead to a severe respiratory illness with 5-12% requiring mechanical ventilation.Standard UK intensive care practice is to consider a tracheostomy after 7-10 days of mechanical ventilation in order to facilitate weaning, reduce duration of mechanical ventilation, shorten intensive care stay and reduce complications relating to prolonged presence of an endotracheal tube. Given the severity of respiratory illness and a mortality in mechanically ventilated COVID 19 patients which exceeds 50%, the benefit of tracheostomy in this group is uncertain.

There are also unique considerations regarding health care professional (HCP) safety when performing tracheostomy in COVID-19 patients due to the potential of aerosol generation and transmission of the infection. ENT UK and other organisations have issued guidance regarding surgical tracheostomy in terms of timing, environment, technique and level of personal protective equipment (PPE). The ability of hospital departments to follow this guidance and the effectiveness of these measures is unknown.

This UK national cohort study aims to assess the effects of tracheostomy in mechanically ventilated COVID-19 patients in terms of the duration of mechanical ventilation, length of ICU and hospital stay and mortality. These data will be related to COVID-19 patients who are mechanically ventilated but do not undergo tracheostomy, as captured by the UK Intensive Care National Audit and Research Centre (ICNARC).

In parallel we will collect data on the tracheostomy procedure itself and compare these to national guidance on tracheostomy in patients diagnosed with COVID-19, and on COVID-19 infections in the surgical and medical teams involved in the tracheostomy procedure.

This proposal builds upon the ongoing COVIDTrach project that has captured data on 550 COVID-19 tracheostomies from 78 NHS hospitals throughout the UK so far. COVIDTrach has successfully brought together surgical, intensive care and anaesthetic specialists to capture early timepoints following tracheostomy. Moving forward, we will work with speech and language therapists and physiotherapists to capture later stages in the patient pathway. This will provide a unique and comprehensive assessment of the role of tracheostomy in COVID-19 patients. It will lay the foundation for further much needed multidisciplinary research into the role of tracheostomy in respiratory disease beyond the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Diagnosed with COVID-19
* Mechanically ventilated
* Undergoing elective surgical or percutaneous tracheostomy
* Health care professionals involved in the tracheostomy procedure (main operator and assistant)

Exclusion Criteria:

* COVID-19 patients undergoing an emergency tracheostomy;
* Patients younger than 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients with COVID-19 who undergo tracheostomy in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 2234 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Time to wean | 12 months
  Clinical outcome in terms of time in days from tracheostomy to successful weaning from mechanical ventilation.

SECONDARY OUTCOMES:
Airway related outcomes | 12 months
  Clinical outcome in terms of length of time from tracheostomy to tracheostomy decannulation.
Complications | 12 months
  Clinical outcome in terms of tracheostomy related complications in terms of bleeding, displaced tube, blocked tube, other.
Length of stay | 12 months
  Clinical outcome in terms of length of stay at intensive care and total length of stay in hospital in days.
Mortality | 12 months
  Clinical outcomes in terms of patient mortality during or following tracheostomy, timing and cause of death
Adherence of tracheostomy procedure to national guidance | 12 months
  Following PPE guidance
Operator wellness | 12 months
  Symptomatic or test positive COVID-19 infection in healthcare professionals involved in the tracheostomy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Nick JI Hamilton, MBChB PhD, Principal Investigator — University College, London
Locations (1):
- University College London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] COVIDTrach collaborative. COVIDTrach: a prospective cohort study of mechanically ventilated patients with COVID-19 undergoing tracheostomy in the UK. BMJ Surg Interv Health Technol. 2021 Jul;3(1):e000077. doi: 10.1136/bmjsit-2020-000077. Epub 2021 Jul 8. PMID 34282409